CLINICAL TRIAL: NCT00463892
Title: A Phase II Study of High-resolution Contrast-enhanced MRI of Regional Lymph Nodes in Patients With Clinically Localized Invasive Melanoma
Brief Title: High-resolution Magnetic Resonance Imaging (MRI) Scans to Look for Spread of Melanoma to Nearby Lymph Nodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Redwood Regional Medical Group (Other)
Responsible Party: Principal Investigator, Peter Brett, M.D., Physician, Redwood Regional Medical Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RRMG #07-001
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Melanoma
Keywords: melanoma; lymph nodes; magnetic resonance imaging; screening; detection
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: High-resolution contrast-enhanced MRI scan — High-resolution contrast-enhanced MRI scan of regional lymph nodes every 6 months on study

SUMMARY:
The study is designed to see if a high-resolution MRI scan of lymph node areas near where a melanoma has been removed from the skin can pick up the spread of melanoma to those lymph nodes with a high degree of accuracy.

DETAILED DESCRIPTION:
When a melanoma of the skin is diagnosed, there is some chance it can spread to nearby lymph nodes, and from there to other parts of the body. Currently, patients with melanoma at low risk for spreading to lymph nodes do not get the lymph nodes assessed except by a physical exam. Those at high risk for spreading to lymph nodes get one or more lymph nodes removed surgically to check for melanoma spread. But physical exam alone will often miss small areas of melanoma in lymph nodes; removal of lymph nodes by surgery is painful and can cause complications. Neither assessment tool is optimal.

This study is designed to see if use of very high-resolution contrast-enhanced MRI scans of lymph node areas near the primary melanoma site in the skin can accurately detect small areas of melanoma spread to those lymph nodes. If this turns out to be the case, in the future, MRI scans could potentially be an alternative for assessing lymph nodes, compared to physical exams alone or surgical removal of the lymph nodes.

In this study, patients with low risk melanoma will receive very high-resolution MRI scans of nearby lymph nodes every 6 months for 5 years of follow-up. If the MRI looks abnormal, the lymph nodes will be biopsied, and results from the biopsy compared to the results from the MRI.

Patients with high risk melanoma will get a baseline MRI of the nearby lymph nodes, and then one or more lymph nodes will be removed (usually by sentinel lymph node biopsy) regardless of the MRI results. Again, results from the biopsy will be compared to the results from the MRI. MRI's will still be repeated every 6 months to assess whether lymph nodes not removed at surgery develop any changes.

We plan to enroll 200 patients on this study and by the end of the study will have a measure of the sensitivity and specificity of high-resolution MRI scans in the detection of melanoma involvement of regional lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* history of invasive cutaneous melanoma stages 1-3 within 2 years of treatment of the melanoma by primary excision
* eligible whether or not a sentinel lymph node biopsy or regional lymph node dissection has been performed
* adequate renal function (creatinine 2 or less)
* life expectancy 2 years of more

Exclusion Criteria:

* history of severe claustrophobia precluding MRI scans
* known hypersensitivity or other contraindication to gadolinium contrast
* known presence of metastatic melanoma at sites beyond regional lymph nodes (stage 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the sensitivity and specificity of high-resolution MRI scans of regional lymph nodes compared to results from regional lymph node biopsy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brett, M.D., Principal Investigator — Redwood Regional Medical Group; David Feinberg, M.D., Ph.D., Principal Investigator — Redwood Regional Medical Group
Locations (1):
- Redwood Regional Medical Group, Sebastopol, California, United States